CLINICAL TRIAL: NCT05470374
Title: Intraoperative Sonographically Guided Resection of Gliomas Not Enhancing Contrast Agent in Magnetic Resonance Imaging: a Randomised, Controlled Trial
Brief Title: Intraoperative Sonographically Guided Resection of Non-enhancing Gliomas
Acronym: SONOGLIO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Neurosurgeon, MD, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non-enhancing Cerebral Gliomas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Glioma extent of resection will be assessed by radiologists blinded for the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound (Experimental): Glioma resection with intraoperative sonography
  Interventions: Procedure: Intraoperative sonography
- Non-ultrasound (No Intervention): Glioma resection without intraoperative sonography

INTERVENTIONS:
Procedure: Intraoperative sonography — ultrasound scanning of brain to search tumor remnants
  Arms: Ultrasound

SUMMARY:
The purpose of the study is to determine whether intraoperative ultrasound guided resection of glioma without contrast enhancement in magnetic resonance imaging can achieve higher extent of resection than surgery without intraoperative sonography

DETAILED DESCRIPTION:
Gliomas, not enhancing contrast agent in magnetic resonance imaging (MRI), are usually low-grade gliomas. They rarely show intraoperative fluorescence using 5-aminolevulinic acid or fluorescein. Intraoperative high-field MRI, sonography and navigation are the only ways to assess extent of their resection during surgery. MRI is the gold standard, but interrupts surgical workflow and only few hospitals are equipped with device like that. Navigation eventually looses it's precision due to brainshift. Ultrasound allows assess tumor remnants in real time but has worse imaging quality. Currently no randomized trials published their results about efficiency of intraoperative sonography in removing low-grade gliomas.

Objective of the study is to determine whether intraoperative ultrasound guided resection of non-enhancing gliomas can achieve higher extent of resection than surgery without intraoperative sonography.

Participants of the study will be randomly operated with and without intraoperative ultrasound. Extent of resection will be assessed in postoperative MRI by blinded radiologists.

ELIGIBILITY:
Inclusion Criteria:

* single supratentorial gliomas without contrast enhancement in preoperative magnetic resonance imaging (presumed low-grade gliomas)
* newly diagnosed
* previously untreated
* Karnofsky Performance Status 60-100%
* age 18-79 years
* performed magnetic resonance imaging with contrast enhancement

Exclusion Criteria:

* glioma spreading to brainstem
* previously performed radiotherapy, chemotherapy or immunotherapy
* planned supratotal tumor resection until neurophysiologically revealed eloquent areas

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Extent of resection in percents | within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100

SECONDARY OUTCOMES:
Gross total resection (Yes or No) | within 48 hours after surgery
  Gross total resection is a total removal of tumor (or 100 percents extent of resection)
Motor function (in grades) | within 10 days after surgery
  Motor function is assessed in Medical Research Council scale
Speech function (in grades) | within 10 days after surgery
  Speech function is assessed in Hendrix scale (2017)
Karnofsky Performance status in percents | within 10 days after surgery
  Assesses patients' possibilities to self-service
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No